CLINICAL TRIAL: NCT01952418
Title: Effect of Video Monitor Size on Adenoma Detection Rate
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Norman Nishioka, MD, Physician, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 2013p001462
Record Dates: First submitted 2013-09-19; First posted 2013-09-30 (Estimated); Results first posted 2017-04-14 (Actual); Last update posted 2017-05-30 (Actual); Status verified 2017-04

CONDITIONS: Colon Adenoma

STUDY DESIGN:
Who Masked: Participant
Masking Description: 15 endoscopists and 1805 patients on which procedures were performed were randomly assigned to each room.
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard monitor (24") (No Intervention): Endoscopists in this arm will perform colonoscopy using the standard size video monitor (24").
- Large monitor (32") (Active Comparator): Subjects randomized to this group will perform colonoscopy while viewing a large video monitor (32").
  Interventions: Device: Monitor size

INTERVENTIONS:
Device: Monitor size — Subjects will be randomized to perform their colonoscopy procedures while viewing a large (32") video monitor or the standard (24") video monitor.
  Arms: Large monitor (32")

SUMMARY:
The goal of this study is to compare the adenoma detection rate achieved while using either a 24" video monitor or a 32" video monitor.

DETAILED DESCRIPTION:
Gastrointestinal endoscopists perfoming routine endoscopic procedures and their patients will be randomized to one of two endoscopy rooms at the MGH Ambulatory Endoscopy Center at Charles River Plaza. The two rooms will have identical equipment with the exception that one room will have the current standard size video monitor (NDS 26") used at this facility while the other room will have a larger video monitor (NDS 32"). The ADR achieved by each physician in each room will be compared.

ELIGIBILITY:
Inclusion Criteria:

* Physician endoscopist performing colonoscopy at Massachusetts General Hospital GI Endoscopy Unit
* Patients receiving these procedures at Massachusetts General Hospital GI Endoscopy Unit

Exclusion Criteria:

* Refusal to participate

Ages: 25 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1805 (Actual)
Dates: Start 2013-10 (Actual); Primary Completion 2014-12 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Norman S Nishioka, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Jovani M, Campbell EJ, Hur C, Joshi AD, Nishioka NS. Effect of video monitor size on polyp detection: a prospective, randomized, controlled trial. Gastrointest Endosc. 2019 Aug;90(2):254-258.e2. doi: 10.1016/j.gie.2019.03.1172. Epub 2019 Apr 12. PMID 30986402

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Standard Monitor (24") | Large Monitor (32")
Started | 910 | 895
Completed | 910 | 895
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: patients who had endoscopy performed in the study
Groups:
- Large Monitor (32"): Endoscopists in this arm will perform colonoscopy using the large size video monitor (32").
- Total: Total of all reporting groups
Arm/Group | Standard Monitor (24") | Large Monitor (32") | Total
Number analyzed (Participants) | 910 | 895 | 1805
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.9 (11.8) | 55.8 (11.5) | 55.3 (11.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 521 | 498 | 1019
  Male | 389 | 397 | 786
Region of Enrollment [Number; unit: participants]
  United States | 910 | 895 | 1805

OUTCOME MEASURES:

1. Primary Outcome: Adenoma Detection Rate (All Indications)
Description: Number of patients with adenoma detected
Time Frame: within 2 weeks (range of 1 day-14 days) of the endoscopy
Population: all indications
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Monitor (24") | Large Monitor (32")
Number analyzed (Participants) | 910 | 895
Participants | 264 | 271

2. Primary Outcome: Adenoma Detection Rate (Screening Exams Only)
Description: Number of patients with adenoma detected
Time Frame: within 2 weeks (range of 1 day-14 days) of the endoscopy
Population: screening exams only
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Monitor (24") | Large Monitor (32")
Number analyzed (Participants) | 491 | 522
Participants | 137 | 157

3. Secondary Outcome: Polyp Detection Rate (All Indications)
Description: Number of patients with polyps detected
Time Frame: recorded during endoscopy (immediate)
Population: all indications
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Monitor (24") | Large Monitor (32")
Number analyzed (Participants) | 910 | 895
Participants | 367 | 424

4. Secondary Outcome: Polyp Detection Rate (Screening Exams Only)
Description: Number of patients with polyps detected
Time Frame: recorded during endoscopy (immediate)
Population: screening exams only
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Monitor (24") | Large Monitor (32")
Number analyzed (Participants) | 491 | 522
Participants | 137 | 157

ADVERSE EVENTS:
Arm/Group | Standard Monitor (24") | Large Monitor (32")
Serious Adverse Events (participants affected / at risk) | 0/910 | 0/895
Other Adverse Events (participants affected / at risk) | 0/910 | 0/895

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes